CLINICAL TRIAL: NCT06952387
Title: Effect of Personalized Blood Pressure Management on Postoperative Complications and Mortality in High-risk Patients Undergoing Major Non-cardiac Surgery: a Randomized Controlled Trial
Brief Title: PeRsonalized Blood prEssure Management on Postoperative Complications and Mortality in hIgh-risk Patients Undergoing Major Non-cardiac Surgery
Acronym: PREMIUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NFEC-2025-134
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hypotension
Keywords: Blood Pressure; Postoperative complications; Mortality; Non-cardiac surgery
MeSH Terms: conditions — Hypotension; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): In patients assigned to control group, clinicians were unaware of the results of preoperative automated 24-h blood pressure monitoring and thus managed blood pressure per institutional routine which generally is to maintain MAP above 60 mmHg. Routine blood pressure management started with the induction of anesthesia and lasted for 2 hours after surgery.
  Interventions: Other: Routine blood pressure management
- Intervention group (Experimental): In patients assigned to intervention group, clinicians were asked to maintain intraoperative MAP above the preoperative baseline MAP (with a maximum MAP target of 110 mmHg and a minimum MAP target of 65mmHg). Personalized blood pressure management started with the induction of anesthesia and lasted for 2 hours after surgery.
  Interventions: Other: Personalized blood pressure management

INTERVENTIONS:
Other: Personalized blood pressure management — In patients assigned to personalized blood pressure management, clinicians were asked to maintain intraoperative MAP at least at the preoperative mean 24-hour MAP (with a maximum MAP target of 110 mmHg) from anesthesia induction to 2 hors after completion of surgery. If the preoperative mean 24-hour MAP was below 65mmHg, intraoperative MAP was maintained at least at 65mmHg.
  The mini fluid challenge (mini-FC, 100ml fluid infusion within 1minute) will be used to assess fluid responsiveness. A positive min-FC response (a stroke volume (SV) increase of at least 5%) will trigger fluid challenge (FC) administration (4ml/kg of balanced crystalloid or colloid within 10 minutes), whereas a negative min-FC response will trigger vasoactive drug administration.
  Other Names: Individualized blood pressure management
  Arms: Intervention group
Other: Routine blood pressure management — In patients assigned to routine blood pressure management, clinicians were blinded to the results of preoperative automated 24-hour blood pressure monitoring, and thus managed blood pressure per institutional routine which generally is to maintain MAP above 60 mmHg.
  The mini fluid challenge (mini-FC, 100ml fluid infusion within 1minute) will be used to assess fluid responsiveness. A positive min-FC response (a stroke volume (SV) increase of at least 5%) will trigger FC administration (4ml/kg of balanced crystalloid or colloid within 10 minutes), whereas a negative min-FC response will trigger vasoactive drug administration.
  Other Names: Standard blood pressure management
  Arms: Control group

SUMMARY:
High-risk populations, particularly elderly individuals and patients with cardiovascular comorbidities, exhibit markedly elevated incidences of postoperative myocardial injury (MINS), acute kidney injury (AKI), and mortality.

Intraoperative hypotension (IOH), a pervasive clinical phenomenon affecting 40%-90% of surgical cases, Substantial observational evidence links IOH severity/duration to ischemic organ injuries (MINS, AKI) and long-term morbidity.Nevertheless, inherent limitations of observational designs-particularly residual confounding-preclude definitive causal inferences. Notably, randomized controlled trials (RCTs) investigating goal-directed hemodynamic interventions demonstrate inconsistent clinical benefits, underscoring the imperative to clarify causal mechanisms between IOH and organ injury. This causal ambiguity arises from two unresolved scientific questions:

(1) Threshold personalization deficit; (2) Therapeutic strategy limitations. In light of current evidence, perioperative hypotension management demands personalized strategies, the investigators propose a multicenter randomized controlled trial (RCT) that aims to clarify the clinical benefits of individualized blood pressure management.

DETAILED DESCRIPTION:
Anesthesia- and surgery-related complications and mortality constitute a critical global public health burden. Annually, over 300 million surgical procedures are performed worldwide, with postoperative complications and mortality standing as predominant contributors to adverse outcomes. High-risk populations, particularly elderly individuals and patients with cardiovascular comorbidities, exhibit markedly elevated incidences of postoperative myocardial injury (MINS), acute kidney injury (AKI), and mortality. Refinement of perioperative management protocols-especially precision-guided hemodynamic control-has emerged as a pivotal strategy for optimizing patient prognosis.

Intraoperative hypotension (IOH), a pervasive clinical phenomenon affecting 40%-90% of surgical cases, is conventionally defined through either absolute thresholds (e.g., systolic blood pressure (SBP) <90 mmHg or mean arterial pressure (MAP) <65 mmHg) or relative reductions from baseline values (>20% decline). Its high prevalence and association with end-organ hypoperfusion have positioned IOH as a central concern in perioperative care. Substantial observational evidence links IOH severity/duration to ischemic organ injuries (MINS, AKI) and long-term morbidity. Nevertheless, inherent limitations of observational designs-particularly residual confounding-preclude definitive causal inferences. Notably, randomized controlled trials (RCTs) investigating goal-directed hemodynamic interventions demonstrate inconsistent clinical benefits, underscoring the imperative to clarify causal mechanisms between IOH and organ injury.

This causal ambiguity arises from two unresolved scientific questions:

1. Threshold personalization deficit: Current paradigms predominantly apply population-based fixed thresholds (e.g., MAP ≥75-80 mmHg vs. ≥60 mmHg), disregarding interindividual hemodynamic variability. Although The Intraoperative Norepinephrine to Control Arterial Pressure (INPRESS) study used personalized blood pressure targets, its approach of measuring baseline blood pressure during a single clinic visit conflicts with current evidence. Research shows that 24-hour ambulatory monitoring is the most reliable method to capture an individual's true baseline blood pressure and daily fluctuations.
2. Therapeutic strategy limitations: Conventional protocols emphasizing aggressive vasopressor use to achieve arbitrary pressure targets may inadvertently increase complications like anastomotic leakage and AKI. Furthermore, the multifactorial etiology of IOH-encompassing hypovolemia, vasoplegia, and impaired cardiac contractility-demands etiology-specific management algorithms rather than universal interventions.

In light of current evidence, perioperative hypotension management demands personalized strategies. To address this need, the investigators propose a multicenter randomized controlled trial (RCT) that pioneers the integration of ambulatory blood pressure monitoring (ABPM) with etiology-specific intervention protocols. This study aims to clarify the clinical benefits of individualized blood pressure management and establish high-quality evidence to advance precision anesthesia practices in perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-90 yr;
* Scheduled to undergo elective non-cardiac major surgery under general anesthesia (with an estimated surgery duration of ≥ 2 hours and an anticipated postoperative hospital stay of ≥ 2 days);
* Patients with high cardiovascular risk, meeting at least one of the following conditions:

  1. History of stroke;
  2. History of coronary artery disease;
  3. History of congestive heart failure;
  4. History of peripheral arterial disease;
  5. Preoperative brain natriuretic peptide (BNP) ≥ 92 mg/L or N-terminal pro-brain natriuretic peptide (NT-proBNP) ≥ 300 ng/L;
  6. Preoperative cardiac troponin (cTn) or high-sensitivity cardiac troponin (hs-cTn) > upper reference limit;
  7. Hypertension requiring medication treatment;
  8. Diabetes requiring medication treatment;
  9. History of chronic kidney disease;
  10. Continuous smoking for 2 years or more, with interruptions of less than one month before the current hospital admission;
  11. Hypercholesterolemia;
  12. History of transient ischemic attack.

Exclusion Criteria:

* Refuse to participate this trial;
* Inability to communicate in the preoperative period because of coma, profound dementia, or language barrier;
* Severe uncontrolled hypertension before surgery (systolic blood pressure ≥ 180 mmHg, diastolic blood pressure ≥ 110 mmHg);
* Severe hepatic dysfunction (Child-Pugh Class C); or severe renal dysfunction required preoperative dialysis; or American Society of Anesthesiologists (ASA) physical status ≥ V; or expectation lifespan ≤ 24h;
* Unstable cardiovascular conditions: acute coronary syndrome, decompensated heart failure, severe arrhythmias, severe valvular heart disease;
* Scheduled to undergo neurosurgical procedures, transplantation, vascular surgery;
* Urgent surgery;
* Diagnosed with sepsis or sepsis shock before surgery.
* Requiring vasopressor treatment before surgery.
* Unable to finish 24-hour automated blood pressure monitor;
* Current participation in another interventional study.
* Any condition deemed ineligible for participation by clinicians.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1624 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
A composite of postoperative complications and mortality within 30 days after surgery | Up to 30 days after surgery
  Defined as a composite of myocardial injury after non-cardiac surgery (MINS), myocardial infarction (MI), postoperative acute heart failure, non-fatal cardiac arrest, stroke, acute kidney injury (AKI), all-cause mortality.

SECONDARY OUTCOMES:
The individual components of the primary composite outcome within 30 days after surgery | Up to 30 days after surgery
  The incidence of individual components of the primary composite outcome (MINS, MI, postoperative acute heart failure, non-fatal cardiac arrest, stroke, AKI and all-cause mortality).
Proportion of ICU admission after surgery | Up to 30 days after surgery
  Proportion of patients admitted in intensive care unit after surgery.
Length of stay in ICU after surgery | Up to 30 days after surgery
  For patients admitted to ICU after surgery, the investigators record the length of stay in the unit.
Length of stay in the hospital after surgery | Up to 30 days after surgery
  Length of stay in the hospital after surgery.
Other major postoperative complications within 30 days after surgery | Up to 30 days after surgery
  Defined as new onset medical events other than primary composite outcome that were deemed harmful and required therapeutic intervention, that is, Grade II or higher on the Clavien-Dindo classification.
Time to first oral intake after surgery | Up to 30 days after surgery
  Defined as the time interval from surgery completion to first oral intake.
Time to first flatus passage after surgery | Up to 30 days after surgery
  Defined as the time interval from surgery completion to first flatus passage

OTHER OUTCOMES:
Overall survival after surgery | Up to 1 year after surgery
  Time from surgery to death
Disability at 6 months after surgery | At 6 months after surgery
  Disability will assessed by 12-item self-administered World Health Organization disability assessment schedule 2.0 (WHODAS 2.0), which covers six domains of functioning with scores from 0 (no difficulty) to 4 (extreme difficulty) and a total score ranging from 0 to 48, with higher scores representing greater disability.
Disability at 1 year after surgery | At 1 year after surgery
  Disability will assessed by 12-item self-administered World Health Organization disability assessment schedule 2.0 (WHODAS 2.0), which covers six domains of functioning with scores from 0 (no difficulty) to 4 (extreme difficulty) and a total score ranging from 0 to 48, with higher scores representing greater disability.
Quality of life at 6 months after surgery | At 6 months after surgery
  Quality of life will assessed by a five-level EuroQol five-dimensional questionnaire (EQ-5D-5L). It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, SelfCare, Usual Activities, Pain/Discomfort, and Anxiety/ Depression. Each dimension has 5 response categories corresponding to no problems, slight problems, moderate problems, severe problems, and unable to do. The instrument is designed for self completion, and respondents also rate their overall health on the day of the interview on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS).
Quality of life at 1 year after surgery | At 1 year after surgery
  Quality of life will assessed by a five-level EuroQol five-dimensional questionnaire (EQ-5D-5L). It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, SelfCare, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response categories corresponding to no problems, slight problems, moderate problems, severe problems, and unable to do. The instrument is designed for self completion, and respondents also rate their overall health on the day of the interview on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Xuan Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (7):
- China (7):
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Panyu Central Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Background] Saugel B, Fletcher N, Gan TJ, Grocott MPW, Myles PS, Sessler DI; PeriOperative Quality Initiative XI (POQI XI) Workgroup Members. PeriOperative Quality Initiative (POQI) international consensus statement on perioperative arterial pressure management. Br J Anaesth. 2024 Aug;133(2):264-276. doi: 10.1016/j.bja.2024.04.046. Epub 2024 Jun 4. PMID 38839472
- [Background] Wanner PM, Wulff DU, Djurdjevic M, Korte W, Schnider TW, Filipovic M. Targeting Higher Intraoperative Blood Pressures Does Not Reduce Adverse Cardiovascular Events Following Noncardiac Surgery. J Am Coll Cardiol. 2021 Nov 2;78(18):1753-1764. doi: 10.1016/j.jacc.2021.08.048. PMID 34711333
- [Background] Marcucci M, Painter TW, Conen D, Lomivorotov V, Sessler DI, Chan MTV, Borges FK, Leslie K, Duceppe E, Martinez-Zapata MJ, Wang CY, Xavier D, Ofori SN, Wang MK, Efremov S, Landoni G, Kleinlugtenbelt YV, Szczeklik W, Schmartz D, Garg AX, Short TG, Wittmann M, Meyhoff CS, Amir M, Torres D, Patel A, Ruetzler K, Parlow JL, Tandon V, Fleischmann E, Polanczyk CA, Lamy A, Jayaram R, Astrakov SV, Wu WKK, Cheong CC, Ayad S, Kirov M, de Nadal M, Likhvantsev VV, Paniagua P, Aguado HJ, Maheshwari K, Whitlock RP, McGillion MH, Vincent J, Copland I, Balasubramanian K, Biccard BM, Srinathan S, Ismoilov S, Pettit S, Stillo D, Kurz A, Belley-Cote EP, Spence J, McIntyre WF, Bangdiwala SI, Guyatt G, Yusuf S, Devereaux PJ; POISE-3 Trial Investigators and Study Groups. Hypotension-Avoidance Versus Hypertension-Avoidance Strategies in Noncardiac Surgery : An International Randomized Controlled Trial. Ann Intern Med. 2023 May;176(5):605-614. doi: 10.7326/M22-3157. Epub 2023 Apr 25. PMID 37094336
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Nicklas JY, Bergholz A, Dake F, Pham HHD, Rabe MC, Schlichting H, Skrovanek S, Flick M, Kouz K, Fischer M, Olotu C, Izbicki JR, Mann O, Fisch M, Schmalfeldt B, Frosch KH, Renne T, Krause L, Zollner C, Saugel B. Personalised blood pressure management during major noncardiac surgery and postoperative neurocognitive disorders: a randomised trial. BJA Open. 2024 Jul 1;11:100294. doi: 10.1016/j.bjao.2024.100294. eCollection 2024 Sep. PMID 39050403
- [Background] Saugel B, Reese PC, Sessler DI, Burfeindt C, Nicklas JY, Pinnschmidt HO, Reuter DA, Sudfeld S. Automated Ambulatory Blood Pressure Measurements and Intraoperative Hypotension in Patients Having Noncardiac Surgery with General Anesthesia: A Prospective Observational Study. Anesthesiology. 2019 Jul;131(1):74-83. doi: 10.1097/ALN.0000000000002703. PMID 30998509